CLINICAL TRIAL: NCT04103021
Title: Effectiveness of Ultrasound Guidance for Port-A-Cath Insertion in Cancer Patients
Brief Title: Ultrasound Guided Port-A-Cath Isertion in Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Omar Mokhtar Hussein (Other)
Responsible Party: Sponsor-Investigator, Omar Mokhtar Hussein, Resident, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ultrasound PAC
Record Dates: First submitted 2019-09-22; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Vascular Access Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Port-a-cath (Experimental): Ultrasound guided Port-a-cath insertion
  Interventions: Device: Port-A-Cath

INTERVENTIONS:
Device: Port-A-Cath — Totally implanted central venous access device

SUMMARY:
Port-A-Cath is a totally implanted central venous access system and one of the most frequently used systems for administration of chemotherapies in oncological patients .

The currently used techniques for placement of totally implantable venous access devices involve the open insertion by cut down technique, or percutaneous puncture of the central vein either by anatomical landmarks or image guided approach by using ultrasound guidance which is increasingly being preferred over the traditional anatomical landmark due to its low complication rate and high technical success rate; as this technique enables the direct visualization of needle entrance and advancement into the target vein

ELIGIBILITY:
Inclusion Criteria:

* cancer patients
* Indicated for receiving long term chemotherapy
* Accepted coagulation profile.

Exclusion Criteria:

* Severe uncorrectable coagulopathy.
* Prior incidence of central vein thrombosis.
* Patients with active infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Early complications | 24 hours
  Early complications associated with Ultrasound guided Port-a-cath insertion periprocedural and within 24 hours

SECONDARY OUTCOMES:
Late complications | Up to 100 months
  complications associated with Ultrasound guided Port-a-cath insertion after 24 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gebauer B, El-Sheik M, Vogt M, Wagner HJ. Combined ultrasound and fluoroscopy guided port catheter implantation--high success and low complication rate. Eur J Radiol. 2009 Mar;69(3):517-22. doi: 10.1016/j.ejrad.2007.10.018. PMID 19340958
- [Background] Mudan S, Giakoustidis A, Morrison D, Iosifidou S, Raobaikady R, Neofytou K, Stebbing J. 1000 Port-A-Cath (R) placements by subclavian vein approach: single surgeon experience. World J Surg. 2015 Feb;39(2):328-34. doi: 10.1007/s00268-014-2802-x. PMID 25245435
- [Background] Granziera E, Scarpa M, Ciccarese A, Filip B, Cagol M, Manfredi V, Alfieri R, Celentano C, Cappellato S, Castoro C, Meroni M. Totally implantable venous access devices: retrospective analysis of different insertion techniques and predictors of complications in 796 devices implanted in a single institution. BMC Surg. 2014 May 8;14:27. doi: 10.1186/1471-2482-14-27. PMID 24886342
- [Background] Capalbo E, Peli M, Lovisatti M, Cosentino M, Ticha V, Cariati M, Cornalba G. Placement of port-a-cath through the right internal jugular vein under ultrasound guidance. Radiol Med. 2013 Jun;118(4):608-15. doi: 10.1007/s11547-012-0894-6. Epub 2012 Oct 22. PMID 23090255
- [Background] Funaki B, Szymski GX, Hackworth CA, Rosenblum JD, Burke R, Chang T, Leef JA. Radiologic placement of subcutaneous infusion chest ports for long-term central venous access. AJR Am J Roentgenol. 1997 Nov;169(5):1431-4. doi: 10.2214/ajr.169.5.9353475.
- [Background] Reeves AR, Seshadri R, Trerotola SO. Recent trends in central venous catheter placement: a comparison of interventional radiology with other specialties. J Vasc Interv Radiol. 2001 Oct;12(10):1211-4. doi: 10.1016/s1051-0443(07)61681-9. PMID 11585888
- [Background] Miccini M, Cassini D, Gregori M, Gazzanelli S, Cassibba S, Biacchi D. Ultrasound-Guided Placement of Central Venous Port Systems via the Right Internal Jugular Vein: Are Chest X-Ray and/or Fluoroscopy Needed to Confirm the Correct Placement of the Device? World J Surg. 2016 Oct;40(10):2353-8. doi: 10.1007/s00268-016-3574-2. PMID 27216807
- [Background] LaRoy JR, White SB, Jayakrishnan T, Dybul S, Ungerer D, Turaga K, Patel PJ. Cost and Morbidity Analysis of Chest Port Insertion: Interventional Radiology Suite Versus Operating Room. J Am Coll Radiol. 2015 Jun;12(6):563-71. doi: 10.1016/j.jacr.2015.01.012. PMID 26047398
- [Background] Kim DH, Ryu DY, Jung HJ, Lee SS. Evaluation of complications of totally implantable central venous port system insertion. Exp Ther Med. 2019 Mar;17(3):2013-2018. doi: 10.3892/etm.2019.7185. Epub 2019 Jan 18. PMID 30867691
- [Background] Cajozzo M, Palumbo VD, Mannino V, Geraci G, Lo Monte AI, Caronia FP, Fatica F, Romano G, Puzhlyakov V, D'Anna R, Cocchiara G. Ultrasound-guided port-a-cath positioning with the new one-shoot technique: thoracic complications. Clin Ter. 2018 Nov-Dec;169(6):e277-e280. doi: 10.7417/CT.2018.2093. PMID 30554248
- [Background] Zaghal A, Khalife M, Mukherji D, El Majzoub N, Shamseddine A, Hoballah J, Marangoni G, Faraj W. Update on totally implantable venous access devices. Surg Oncol. 2012 Sep;21(3):207-15. doi: 10.1016/j.suronc.2012.02.003. Epub 2012 Mar 17. PMID 22425356